CLINICAL TRIAL: NCT04009135
Title: The Internet Therapy for Depression Trial (INTEREST): A Doubly-randomized, Patient-preference, Controlled Feasibility Trial Comparing iACT, iCBT, and Attention Control
Brief Title: The Internet Therapy for Depression Trial
Acronym: INTEREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Joshua Rash, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HREB2018.275
Record Dates: First submitted 2019-06-17; First posted 2019-07-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain; Major Depressive Disorder
Keywords: Chronic non-cancer pain; Major depression; Internet therapies; Cognitive behaviour therapy; Acceptance and commitment therapy
MeSH Terms: conditions — Chronic Pain; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Doubly-randomized, patient-preference trial with two active study interventions and one control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A research assistant not affiliated with the study will use Research Randomizer (http://www.randomizer.org/) to generate lists of randomly sequenced numbers to allocate patients to trial arm. To reduce biases and expectation effects, the research assistant will not be aware of what condition the patients are allocated when conducting baseline assessments and a research assistant not affiliated with the research will complete outcome assessments without being aware of allocation. Interventionists will be aware of which group patients are allocated to, as will patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- internet delivered cognitive behavioural therapy (iCBT) (Experimental): The intervention comprises 7 weekly online modules available through Therapist Assisted Online (TAO), including: 1) psychoeducation about chronic pain and depression; 2) thoughts and feelings; 3) understanding stress and relaxation; 4) unhealthy and healthy thoughts; 5) layers of thinking; 6) core beliefs; and 7) relationship, lifestyle, problem solving, and relapse prevention. Online content is supplemented with weekly coaching sessions performed via video-conference with doctoral students of Clinical Psychology.
  Interventions: Behavioral: internet delivered cognitive behavioural therapy (iCBT)
- online delivered acceptance and commitment therapy (iACT) (Experimental): The intervention comprises 7 weekly online modules available through Therapist Assisted Online (TAO), including: 1) psychoeducation about chronic pain and depression; 2) introduction to ACT; 3) cognitive fusion and defusion; 4) thinking mind versus observing mind & acceptance; 5) mindfulness; 6) values; and 7) taking action. Online content is supplemented with weekly coaching sessions performed via video-conference with doctoral students of Clinical Psychology.
  Interventions: Behavioral: online delivered acceptance and commitment therapy (iACT)
- Attention Control (AC) (Placebo Comparator): Patients in the control condition will be given access online psychoeducation about depression and chronic pain. They will be provided weekly phone calls to query symptoms and well-being.
  Interventions: Other: Attention Control (AC)

INTERVENTIONS:
Behavioral: internet delivered cognitive behavioural therapy (iCBT) — The intervention comprises 7 weekly online modules available through Therapist Assisted Online (TAO), including: 1) psychoeducation about chronic pain and depression; 2) thoughts and feelings; 3) understanding stress and relaxation; 4) unhealthy and healthy thoughts; 5) layers of thinking; 6) core beliefs; and 7) relationship, lifestyle, problem solving, and relapse prevention. Online content is supplemented with weekly coaching sessions performed via video-conference with doctoral students of Clinical Psychology.
  Arms: internet delivered cognitive behavioural therapy (iCBT)
Behavioral: online delivered acceptance and commitment therapy (iACT) — The intervention comprises 7 weekly online modules available through Therapist Assisted Online (TAO), including: 1) psychoeducation about chronic pain and depression; 2) introduction to ACT; 3) cognitive fusion and defusion; 4) thinking mind versus observing mind & acceptance; 5) mindfulness; 6) values; and 7) taking action. Online content is supplemented with weekly coaching sessions performed via video-conference with doctoral students of Clinical Psychology.
  Arms: online delivered acceptance and commitment therapy (iACT)
Other: Attention Control (AC) — 1-module of psychoeducation about chronic pain and major depression. Weekly contact to complete measures of symptomatology and well-being.
  Arms: Attention Control (AC)

SUMMARY:
The objective of this trial is to collect data on the feasibility, acceptability, and preliminary effectiveness of internet delivered Cognitive Beaviour Therapy (iCBT) and Acceptance and Commitment Therapy (iACT) interventions tailored towards the treatment of depression and chronic pain using a doubly-randomized, attention-controlled, non-blinded, patient-preference design.

DETAILED DESCRIPTION:
The primary objective is to collect data on the feasibility, acceptability, and preliminary effectiveness of internet delivered Cognitive Beaviour Therapy (iCBT) and Acceptance and Commitment Therapy (iACT) on depressed mood among individuals with chronic pain relative to attention control (AC). The secondary objectives are to evaluate the efficacy of iCBT and iACT on clinically relevant outcomes endorsed by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT). Adults with chronic non-cancer pain and major depression will be randomized to receive iACT, iCBT, or AC. The interventions comprise 7 weekly online modules available through Therapist Assisted Online (TAO). Patients will be contacted weekly by a member of the study team who will be acting as their personalized "online therapy coach."

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* 18 years of age or older
* have a primary diagnosis of chronic non-cancer pain.
* meet DSM-5 criteria for a diagnosis of major depressive disorder
* have access to the internet, email, and telephone
* can commit to the demands and timelines of the trial.
* Given high comorbidity in this population, patients with sleep disturbance or comorbid anxiety will also be eligible to participate.

Exclusion Criteria:

* diagnosis of cognitive impairment (e.g., dementia)
* active suicidal ideation
* severe psychopathology (e.g., schizophrenia)
* unable to sign a safety contract for the duration of the trial
* concurrent participation in psychotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Screening and Consent Rates | Through study completion, up to 2-years
  The number of patients with CNCP and suspected major depression who are referred for screening will be recorded. Eligibility rate will be calculated as the number of patients who meet full inclusion criteria divided by the number of patients referred for screening. Number of patients declining referral for screening and reasons for exclusion will be documented. Consent rate will be calculated by dividing the number of patients who consent to undergoing randomization by the number who met full inclusion criteria.
Change in symptoms of depression measured using the Patient Health Questionnaire - 9 (PHQ-9) | Change from baseline to end of treatment (i.e., week 8).
  Change in symptoms of depression as measured using the PHQ-9 from baseline to post-intervention. Scores range from 0-27 with higher scores reflecting greater symptoms of depressed mood.
Adherence to intervention measured as frequency of visits to online modules. | End of treatment (i.e., week 8)
  Intervention adherence will be measured using data recorded by Therapist Assisted Online (TAO) program and include: 1) frequency of visits to TAO modules throughout weeks 1 to 8.
Perceived acceptability of treatment measured using qualitative interviews | Completion of the intervention (i.e., week 8)
  Acceptability data will be collected using semi-structured interviews with patients. Open ended questions will be asked to ascertain the following: 1) acceptability of the delivered intervention; 2) perceived value, benefits, harms and unintended consequences of the delivered intervention; 3) perceived need for refinement of the delivered intervention.

SECONDARY OUTCOMES:
Change in physical function measured using the pain interference subscale of the Brief Pain Inventory - Short Form (BPI-SF) | Baseline, 4-weeks, and post-intervention (i.e., week 8)
  Change in pain interference between baseline and post-intervention will be measured using the Brief Pain Inventory - Short Form (BPI-SF). Pain interference is measured s the average degree to which pain impacts seven daily activities (e.g., activity, work, sleep). Scores range from 0 to 10 with higher scores reflecting greater pain-related interference.
Change in emotion function measured using the Depression, Anxiety Stress Scale - 21 (DASS-21). | Baseline and through study completion, an average of 8-weeks.
  Change in depression, anxiety and stress between baseline and post-intervention measured using the Depression, Anxiety Stress Scale - 21 (DASS-21). The DASS is a 21-item Likert scale with questions ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The 21 questions are divided into three scales, each comprising of 7 questions: depression, anxiety, and stress. Scores for each subscale range between 0 and 21 with higher scores reflecting greater levels of depression, anxiety, and stress.
Change in pain severity will be measured using the pain severity composite scale of the Brief Pain Inventory - Short Form (BPI-SF) | Baseline and through study completion, an average of 8-weeks.
  Change in pain severity between baseline and post-intervention will be measured using the pain severity composite of the Brief Pain Inventory - Short Form (BPI-SF). Pain severity is measured using the average rating of pain made across the previous 24-hour period (e.g., average pain, worst pain, least pain). Scores range from 0 to 10 with higher scores reflecting greater pain severity.
Change in psychological flexibility measured using the Multidimensional Psychological Flexibility Inventory (MPFI). | Baseline and through study completion, an average of 8-weeks.
  Change in psychological flexibility between baseline and post-intervention measured using the Multidimensional Psychological Flexibility Inventory (MPFI). The MPFI is a 60-item scale measuring 6 dimensions of psychological flexibility and 6 dimensions of psychological inflexibility as posited by the Hexaflex model. Each item is rated on a 6-point scale ranging from 1 (never or never true) to 6 (always or always true). Measures of psychological flexibility and inflexibility are calculated as the average score across the subscales representing each dimension. Scores range from 1 to 6 with higher scores representing higher levels of the dimensions being assessed.
Mediators of change for cognitive behavioural therapy measured using change in the cognitive behavioural therapy skills questionnaire. | Baseline and through study completion, an average of 8-weeks.
  Change in cognitive behavioural therapy (CBT) skill utilization among patients allocated to the CBT group will be measured among patients assigned to the CBT group using the CBT skills questionnaire. The CBT skills questionnaire is a 16-item self-report measure that assesses the client's frequency and performance of CBT utilization. It is a 5-point Likert scale ranging from 1 ("I don't do this") to 5 ("I always do this"). Higher scores reflect greater utilization of CBT skills.
Mediators of change for acceptance and commitment therapy measured using change in the acceptance and action questionnaire. | Baseline and through study completion, an average of 8-weeks.
  Change in acceptance of chronic pain will be measured among patients assigned to the acceptance and commitment therapy (ACT) group using the Acceptance and Action Questionnaire (AAQ-II). The AAQ-II is a 7-item self-report measure. Patients rate how true statements are to them on a scale of 1 (never true) to 7 (always true). Score ranges from 7-49, with higher scores reflecting less acceptance and commitment.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bell LV, Cornish P, Flusk D, Garland SN, Rash JA. The INternet ThERapy for deprESsion Trial (INTEREST): protocol for a patient-preference, randomised controlled feasibility trial comparing iACT, iCBT and attention control among individuals with comorbid chronic pain and depression. BMJ Open. 2020 Feb 28;10(2):e033350. doi: 10.1136/bmjopen-2019-033350. PMID 32114466